CLINICAL TRIAL: NCT00585234
Title: Tools for Objective Clinical Assessment of Pediatric Spinal Deformity and the Results of Surgical Intervention--Simultaneous Measurement of Sagittal and Coronal Balance and Symmetry With Digital Photography.
Brief Title: Tools for the Objective Clinical Assessment of Pediatric Spinal Deformity
Status: Withdrawn | Type: Observational
Why Stopped: Study has been withdrawn.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, john t. smith, Clinical Professor, University of Utah
Other Study IDs: 00014137; IRB# 00014137
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Thoracic Insufficiency Syndrome; TIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: We intend to photograph male and female subjects from age 1 through skeletal maturity. Healthy children will be photographed to determine the normative characteristics of thoracic function using this technique. We will also enroll patients with thoracic pathology to determine how digital imaging can document thoracic dysfunction. There are no specific disease related exclusion criteria. Participation is voluntary.
  Interventions: Other: Digital Photography

INTERVENTIONS:
Other: Digital Photography — Digital Photography

SUMMARY:
This project seeks to develop a standardized technique for simultaneous capturing bi-planar images of patients against a standard background with a grid that can be used later for the quantitative determination of global balance and thoracic symmetry.

We hypothesize that patients who are successfully managed with surgery will demonstrate an improvement in global balance and thoracic symmetry that can be accurately measured. This measurement station will be specifically developed to provide a standardized, reproducible means to compare clinical assessments of surgical and non-surgical outcomes, and establish normative data for comparison. This standardized tool can be established at multiple centers for use in multicenter trials.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants from 1- skeletal maturity

Exclusion Criteria:

* no specific disease related exclusion criteria

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary Care Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Improvement in overall global balance following surgical intervention | Dec 2005-Dec 2008

SECONDARY OUTCOMES:
Improvement in overall global balance | Dec 2005-Dec 2008

CONTACTS AND LOCATIONS:
Overall Officials: John T Smith, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States